CLINICAL TRIAL: NCT00727584
Title: SCORAD: A Randomised Feasibility Study of Single Fraction Radiotherapy Compared to Multi-fraction Radiotherapy in Patients With Metastatic Spinal Cord Compression
Brief Title: Radiation Therapy in Treating Patients With Metastatic Spinal Cord Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000599886; CRUK-UCL-BRD-07-010; CRUK-SCORAD; ISRCTN97555949; EU-20863
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Spinal Cord Compression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: spinal cord compression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Spinal Cord Compression | interventions — Radiotherapy

ARMS (2):
- Arm I (multi-fraction radiotherapy) (Active Comparator): Patients undergo 5 fractions of 20 Gy external-beam radiotherapy.
  Interventions: Radiation: radiation therapy
- Arm II (single-fraction radiotherapy) (Experimental): Patients undergo 1 fraction of 8 Gy external beam radiotherapy.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Patients undergo external beam radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known which radiation therapy regimen is more effective in treating metastatic spinal cord compression.

PURPOSE: This randomized clinical trial is comparing two radiation therapy regimens to see how well they work in treating patients with metastatic spinal cord compression.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine whether a phase III randomized study comparing a single-fraction of radiotherapy with multi-fraction radiotherapy is acceptable to clinicians and to patients with metastatic spinal cord compression.
* To determine the feasibility of conducting this study in the United Kingdom.

OUTLINE: This is a multicenter study. Patients are stratified by treatment center and known prognostic factors (ambulatory status at diagnosis, primary tumor type, and extent of disease [spinal metastases only vs spinal and non-bony metastases]). Patients are randomized to 1 of 2 treatment arms.

* Arm I (multi-fraction radiotherapy): Patients undergo 5 fractions of 20 Gy external-beam radiotherapy.
* Arm II (single-fraction radiotherapy): Patients undergo 1 fraction of 8 Gy external beam radiotherapy.

Patients undergo assessment of ambulatory status, quality of life, bladder and bowel function, and acute toxicity via self-reported questionnaires and telephone follow-ups at baseline and weeks 1, 4, 8, and 12.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant disease
* Proven diagnosis of metastatic spinal cord compression on MRI or CT scan

  * Single site of compression OR multiple sites that can be treated within a single radiation treatment field
* No patient for whom surgery or chemotherapy treatment is more appropriate
* No multiple myeloma as primary cancer

PATIENT CHARACTERISTICS:

* Life expectancy > 1 month
* Not pregnant
* Willing and able to complete assessment forms
* Able to give informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Patient accrual per center over a 12-month period

SECONDARY OUTCOMES:
Ambulatory status at 1, 4, 8, and 12 weeks from day 1 of treatment compared to baseline
Bladder and bowel function at 1, 4, 8, and 12 weeks from day 1 of treatment compared to baseline
Acute side effects using RTOG scales at 1, 4, 8, and 12 weeks from day 1 of treatment
Quality of life as measured by the EORTC QLQ-C30 questionnaire at 1, 4, 8, and 12 weeks from day 1 of treatment compared to baseline
Further treatment
Overall survival at 3, 6, and 12 months
Total number of days spent in hospital
Preferred place of care
Number of patients eligible but not randomized and reasons for non-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Hoskin, MD, Principal Investigator — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (4):
- United Kingdom (4):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Cancer Research UK and University College London Cancer Trials Centre, Northwood, England
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Christie Hospital, Manchester